CLINICAL TRIAL: NCT00469495
Title: Empiric Antihelminthic Therapy Combined With Antimony in the Treatment of Cutaneous Leishmaniasis: A Randomized Controlled Trial in Subjects Co-Infected With Helminths and Leishmania Brasiliensis
Brief Title: Antihelminthic Therapy Combined With Antimony in the Treatment of Cutaneous Leishmaniasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitário Professor Edgard Santos (Other)
Responsible Party: Edgar M. Carvalho, Universidade Federal da Bahia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0701008939
Record Dates: First submitted 2007-05-02; First posted 2007-05-04 (Estimated); Last update posted 2009-08-26 (Estimated); Status verified 2009-08

CONDITIONS: Leishmaniasis, Cutaneous; Helminthiasis
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Helminthiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Anti-helminthic
Drug: meglumine antimony

SUMMARY:
The purpose of this project is to investigate the efficacy of early, empiric anti-helminthic therapy combined with standard pentavalent antimony in the treatment of subjects co-infected with helminths and cutaneous leishmaniasis caused by L. brasiliensis. The study hypothesis is that early intervention with antihelminthic therapy will improve response rates to antimony in subjects with cutaneous leishmaniasis.

DETAILED DESCRIPTION:
Leishmaniases are a group of diseases caused by a parasite and transmitted by the sand fly. There are a number of diseases associated with infection ranging from simple skin lesions to a severe, fatal form. The standard treatment of cutaneous leishmaniasis (CL) is a 20 day course of antimony which, although fairly effective, has multiple side effects and is difficult to administer. The populations that are affected by leishmaniasis are usually also affected by intestinal helminths (worms). It is unknown what effect these two diseases have on each other and the immune system. As pathology in CL is mediated by an inflammatory reaction and helminths down regulate inflammation, helminthic infection may be beneficial for leishmaniasis. However, a recent study by our research group suggested that subjects infected with both leishmania and helminths have longer healing times and are less likely to respond to antimony. Since failure of initial therapy often results in repeat courses of the drug or development of more severe disease, we propose a study to investigate the role of early treatment for co-existing helminth infections in improving response rates to antimony in subjects with CL.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of CL based on the presence of typical skin lesions and a positive Montenegro skin test
* Evidence of helminthic infection by parasitological examination of first stool sample
* Males or females between 13 and 50 years of age
* Maximum of 3 ulcers with no more than 2 body regions involved
* Period of 15 to 60 days from the onset of the first ulcer
* Subject agreement to follow-up visits and therapy
* Ability to give informed consent

Exclusion Criteria:

* Pregnancy
* Breastfeeding mothers
* Presence of mucosal disease
* History of prior treatment with antimonial drugs.
* History of prior treatment with anthelminthic drugs within the last 6 months.
* History of allergy to pentavalent antimony or antihelminthic
* Presence of underlying disease which affects the immune response, such as HIV and diabetes mellitus

Ages: 13 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Bidirectional measurements will be taken of the subjects' lesions at each visit and will be categorized as active or healed by a dermatologist. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Edgar M Carvalho, MD, Principal Investigator — Federal University of Bahia
Locations (1):
- Posto de Saude de Corte de Pedra, Salvador, Estado de Bahia, Brazil

REFERENCES:
- [Derived] Newlove T, Guimaraes LH, Morgan DJ, Alcantara L, Glesby MJ, Carvalho EM, Machado PR. Antihelminthic therapy and antimony in cutaneous leishmaniasis: a randomized, double-blind, placebo-controlled trial in patients co-infected with helminths and Leishmania braziliensis. Am J Trop Med Hyg. 2011 Apr;84(4):551-5. doi: 10.4269/ajtmh.2011.10-0423. PMID 21460008